CLINICAL TRIAL: NCT01647191
Title: Reducing Hepatitis C Virus (HCV)/Human Immunodeficient Virus (HIV) Risk Behaviors Among Injection Drug Users in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JDu-001
Record Dates: First submitted 2012-04-17; First posted 2012-07-23 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2012-07

CONDITIONS: Hepatitis C
Keywords: HCV，; drug users，; intervention
MeSH Terms: conditions — Hepatitis C; Drug Misuse | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): The investigators will use a variety of learning techniques, including lecture, brainstorming, small and large group activity, individual worksheets, role-play, and video player. For example, small teams of up to 5 participants will conduct role-plays; large groups also will be assembled to encourage talking about HCV-related risk reduction behavior.
  Interventions: Behavioral: intervention group
- control group (Active Comparator): The investigators will adopt previous treatment in the clinics to intervent the patients without any type of target intervention for this group.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: intervention group — The investigators will use a variety of learning techniques, including lecture, brainstorming, small and large group activity, individual worksheets, role-play, and video player. For example, small teams of up to 5 participants will conduct role-plays; large groups also will be assembled to encourage talking about HCV-related risk reduction behavior.
  Other Names: some types intervention activities for this group
  Arms: intervention group
Behavioral: control group — The investigators will adopt previous treatment in the clinics to intervent the patients
  Other Names: without any type of target intervention for this group
  Arms: control group

SUMMARY:
The proposed study will investigate the knowledge level, attitudes, and perceptions among staff of Methadone Maintenance Treatment (MMT) clinics and intravenous drug users (IDUs) who attending MMT clinics, which is the most reachable population for HCV/HIV intervention in China. This study will also explore the barriers that prevent IDUs from getting HCV/HIV intervention/prevention and medical care services. This study will help to understand and address this important problem in China and other Asian countries.

DETAILED DESCRIPTION:
The investigators propose to conduct 3 inter-related studies over 4 years using both qualitative and quantitative research methods to address a series of research questions. Firstly, The investigators will begin by assessing HCV/HIV knowledge, attitudes, perceptions, risk behaviors, and infection among IDUs in MMT clinics (Study 1) and HCV/HIV knowledge, attitudes, and HCV/HIV-related services among MMT staff (Study 2). Secondly, based on knowledge accumulated from Studies 1 & 2; The investigators will adapt and develop HCV/HIV education materials appropriate for Chinese IDUs and drug treatment service providers, and then use the Transtheoretical Model of Behavior Change as a conceptual model to measure if our educational program will increase patients' readiness to consider changing HCV/HIV risk behaviors and getting medical care for HCV/HIV (Study 3). Finally, by integrating findings of these three studies and by consulting with leading experts in HCV/HIV. The investigators plan to develop HCV/HIV intervention program applicable in China, which can be tested in future formal experimental trials.

ELIGIBILITY:
Inclusion Criteria:

* several failed attempts to quit the use of heroin
* at least two terms in a detoxification center
* age at least 20 years
* being a registered local resident of the area in which the clinic is located
* being of good civil character

Exclusion Criteria:

* there is no exclusion criteria

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Knowledge、Risk Behaviors and some other aspects related to HCV/HIV will be measured among IDUs in MMT | 3 months
  HCV/HIV knowledge, attitudes, perceptions, risk behaviors, and infections (HIV, HCV, and HIV/HCV co-infection) will be measured by HCV/HIV knowledge questionnaire,HCV/HIV self-efficacy scale,Attitudes and practices regarding HCV/HIV infection among IDUs in MMT

SECONDARY OUTCOMES:
The barriers will be measured. | 3 months
  The barriers that impact IDUs receiving HCV/HIV-related intervention and medical service will be measured by Focus group instruments,which including potential topics as follow: what kind of HCV/HIV service do you provide to IDUs? What are the most important barriers that impact IDUs obtaining HCV services? What are the important barriers that prevent you from offering HCV/HIV-related service to IDUs? What recommendation do you have to increase HCV/HIV-related medical services in MMT clinics?.
The ways will be measured. | 3 months
  The ways to facilitate MMT staff to provide HCV/HIV-related services to IDUs will be measured by HCV/HIV self-efficacy scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, M.D, Principal Investigator — Shanghai Mental Health Center
Locations (2):
- China (2):
  - Shanghai Hong Kou MMT clinic, Shanghai, Shanghai Municipality
  - Shanghai Yang Pu MMT clinic, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhang JY, Li ZB, Zhang L, Wang J, Huang LP, Zhan GL, Li Z, Du J, Zhao M. DOES IT WORK? -a randomized controlled trial to test the efficacy of HCV and HIV-related education on drug users in MMT, China. BMC Infect Dis. 2019 Sep 5;19(1):774. doi: 10.1186/s12879-019-4421-5. PMID 31488064
- [Derived] Li ZB, Zhang L, Wang J, Huang LP, Zhou ZR, Cao YN, Zhao M, Du J. Hepatitis C infection, related services, and barriers to HCV treatment among drug users in methadone maintenance treatment (MMT) clinics in Shanghai, China. Harm Reduct J. 2017 Nov 2;14(1):71. doi: 10.1186/s12954-017-0197-3. PMID 29096647